CLINICAL TRIAL: NCT02069106
Title: An 8-Week, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Daily Pro-Omega LDL for Low-Density Lipoprotein Cholesterol and Triglyceride Reduction in Subjects With Mixed Hyperlipoproteinemia
Brief Title: Efficacy Study of Daily Pro-Omega LDL for Low-Density Lipoprotein Cholesterol and Triglyceride Reduction
Acronym: PrOteCT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Nordic Pharma, USA (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1001-PR-003-09092013
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Mixed Hyperlipoproteinemia
Keywords: low density lipoprotein cholesterol; triglycerides; mixed hyperlipoproteinemia; Dehydroascorbic Acid; Eicosapentaenoic Acid; Fish oil
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pro-Omega LDL (Experimental): 3 capsules 1000 mg BID for 8 weeks
  Interventions: Dietary Supplement: Pro-Omega LDL
- Placebo (Placebo Comparator): 3 capsules BID for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Pro-Omega LDL
  Arms: Pro-Omega LDL
Other: Placebo
  Arms: Placebo

SUMMARY:
Pro-Omega LDL reduces low-density lipoprotein cholesterol and triglycerides in subjects with mixed hyperlipoproteinemia.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, ≥18 years of age.
* History (>3months) of LDL-C ≥130 mg/dl to ≤190 mg/dL
* Triglycerides (TG) > 200 to <750 mg/dL
* Able to understand and cooperate with study procedures, and have signed a written informed consent prior to any study procedures.
* Willing to maintain a stable diet and level of activity throughout the trial. Willing to maintain current activity level and diet throughout the trial.
* If, of childbearing age, must be on a medically approved form of birth control as identified by the investigator in this trial
* History (> 3 months) of taking a statin medication (HMG-CoA reductase inhibitor, including Lipitor, Zocor, Crestor, Pravachol, Lescol, Livalo) without problems, and would be willing to withdraw from statin for the duration of the trial (4 weeks without statin prior to randomization for washout period, then treatment with protocol medication for 10 week duration of the trial)

Exclusion Criteria:

* Individuals with intolerance of, or allergy to red yeast rice or omega 3 fatty acids.
* Individuals currently taking a statin (HMG-CoA Reductase inhibitor) including Lipitor, Zocor, Crestor, Pravachol, Lescol, Livalo) or other lipid metabolism altering product within four (4) weeks prior to randomization who do not wish to withdraw from therapy.
* Individual taking prescription or over the counter medications (including dietary supplements) known to alter lipid metabolism within four (4) weeks of randomization. Medications excluded within 4 weeks of randomization are: prescription omega-3 fatty acids, statins, bile acid sequestrants, cholesterol absorption inhibitors, niacin or fibrates. Dietary supplements excluded within 4 weeks prior to randomization are: L-carnitine, policosanol, guggulipid, sterol/stanol products, red rice yeast supplements, garlic supplements, soy isoflavone supplements, niacin or its analogues, probiotics and dietary fiber supplements (including >2 teaspoons Metamucil or psyllium-containing supplements per day and prebiotics), or any dietary supplement or vitamin complex product containing omega 3 acids or fish oil.
* Use of systemic corticosteroids, androgens (except androgens for hypogonadism to restore normal levels), phenytoin, erythromycin and other macrolides, and thyroid hormones (except stable-dose thyroid replacement therapy for four (4) weeks prior to enrollment).
* Use of the anticoagulants warfarin (Coumadin) or dabigatran (Pradaxa), apixaban (Eliquis) or rivaroxaban (Xarelto).
* Pregnant or lactating women, or women of childbearing potential who are not complying with an approved method of contraception. A woman is considered to be of childbearing potential unless she is post-hysterectomy, one or more years postmenopausal, or one or more years post-tubal ligation.
* Individuals with a history of myopathy, defined as a creatine phosphokinase (CPK) >450 U/L and/or unexplained muscle pain on statins.
* Type I or type II diabetes mellitus or HbA1c ≥7.0%
* History of significant cardiovascular or coronary heart disease (CVD or CHD) as defined by having had a coronary artery bypass procedure, coronary stent or angioplasty, or myocardial infarction.
* Current or recent (within six months) history of significant gastrointestinal, renal, pulmonary, hepatic or biliary disease
* History of cancer, other than non-melanoma skin cancer and basal cell carcinoma, within the previous five years.
* Poorly controlled or uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥95 mm Hg).
* Recent history (within past 6 months) of excessive alcohol use, defined as >14 drinks per week (One drink = 12 oz. beer, 4 oz. wine, 1.5 oz. hard liquor).
* Exposure to any investigational agent within 4 weeks prior to Visit 1.
* Has a condition the Investigator believes would interfere with the evaluation of the subject, or may put the subject at undue risk during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Low-density lipoprotein cholesterol (LDL-C) | 8 weeks
Triglycerides (TG) | 8 weeks

SECONDARY OUTCOMES:
Total cholesterol | 8 weeks
High-density lipoprotein cholesterol (HDL-C) | 8 weeks
non-HDL-C | 8 weeks
LDL-C/HDL-C ratio | 8 weeks
C-reactive protein | 8 weeks
Adverse events | 4 and 8 weeks
Offset effect | 2 weeks after withdrawal
  Offset effect of Pro-Omega LDL two weeks after withdrawal of placebo and Pro-Omega LDL on serum markers

CONTACTS AND LOCATIONS:
Overall Officials: David Becker, MD, Principal Investigator — Chestnut Hill Temple Cardiology